CLINICAL TRIAL: NCT04896151
Title: Assessing the Utility of MMPI-2-RF-EX in Detecting Simulated Underreporting of Current Suicide Risk in Military Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Minnesota (Other); Rutgers University (Other)
Responsible Party: Principal Investigator, Lauren Khazem, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020B0414
Record Dates: First submitted 2021-05-01; First posted 2021-05-21 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Suicidal Ideation; Suicidal
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MMPI (Active Comparator): Participants will be instructed to complete the MMPI-2-RF-EX and other measures under standard conditions (e.g., to not simulate underreporting of suicide risk).
  Interventions: Diagnostic Test: Minnesota Multiphasic Personality Inventory -2- Restructured Form - Experimental
- Simulation MMPI (Experimental): Participants will be instructed to conceal current suicide risk when completing the MMPI-2-RF-EX and other measures.
  Interventions: Diagnostic Test: Minnesota Multiphasic Personality Inventory -2- Restructured Form - Experimental

INTERVENTIONS:
Diagnostic Test: Minnesota Multiphasic Personality Inventory -2- Restructured Form - Experimental — The MMPI-2-RF-EX is a broadband, self-report measure of personality and psychopathology was developed for research purposes in order to develop the MMPI-3 (Ben-Porath & Tellegen, 2020), which is comprised of a subset of MMPI-2-RF-EX items.
  Other Names: MMPI-2-RF-EX

SUMMARY:
The aim of the current project are is examine the incremental predictive utility of the MMPI-2-RF-EX validity scales in detecting simulated underreporting of suicide risk on the MMPI-2-RF-EX and other self-report measures of suicide risk in 150 military Veterans experiencing past-month death or suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* US military veteran
* death or suicidal ideation/suicide attempt within the past month

Exclusion Criteria:

* non-Veteran status
* acute intoxication or active psychosis precluding provision of informed consent
* an inability to communicate and comprehend English
* residence outside the United States
* lack of past-month death/suicide ideation or attempt
* younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
MMPI-2-RF-EX Suicidal/Death Ideation scale | Baseline
  The MMPI-2-RF-EX Suicidal/Death Ideation scale is a self-report measure of current suicide risk contained within the instrument. T scores range from 45 to 100, with higher scores indicative of greater suicide risk.
Beck Scale for Suicide Ideation (BSS) | Baseline
  The BSS is a 21-item measure of past-week suicide ideation and desire for death. Responses to items are scored on a 3-point Likert scale (range of 0- 2). Scores range from 0 to 42, with higher scores indicating greater suicide risk.

SECONDARY OUTCOMES:
Suicide Cognitions Scale (SCS) | Baseline
  The SCS is an 18-item survey measuring suicide-related thoughts and beliefs, unclouding hopelessness, perceived burdensomeness, entrapment, and unbearability. Respondents rate their agreement with each statement on a 5-point Likert scale. Scores range from 18-90, with higher scores indicating more severe suicide risk.

OTHER OUTCOMES:
Short Grit Scale | Baseline
  The Short Grit Scale is an 8-item measure of trait-level perseverance and passion for long-term goals. Possible scores range from 5 to 40, with higher scores indicting higher levels of grit.
MMPI Posttest Inquiry (PTI) | Baseline
  The PTI assesses participants' compliance with condition-specific instructions for completing the MMPI and was adapted for the proposed research
PTSD Checklist for DSM-5 (PCL-5) PTSD Checklist for DSM-5 | Baseline
  The PCL-5 is a self-report measure assessing the severity of 20 PTSD symptoms. Scores range from 0 to 80, with higher scores indicating greater PTSD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Khazem, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khazem LR, Keen MA, Rodriguez TR, Ingram PB, Hay JM, Long CM, Bryan CJ, Anestis JC. Detecting Simulated Underreporting on the Minnesota Multiphasic Personality Inventory-3 (MMPI-3) in Veterans With Past-Month Death/Suicide Ideation. Suicide Life Threat Behav. 2025 Apr;55(2):e13170. doi: 10.1111/sltb.13170. PMID 40135882

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04896151/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT04896151/ICF_001.pdf